CLINICAL TRIAL: NCT03273881
Title: Effect of Intrapartum Glucose With Compared to Without Constant Intravenous Insulin on Neonatal Hypoglycemia Among Diabetic Women. A Randomized Controlled Trial
Brief Title: Intrapartum Glucose and Insulin Compared to Glucose Alone in Diabetic Women
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: HaEmek Medical Center, Israel (Other)
Collaborators: Holy Family Hospital, Nazareth, Israel (Other)
Responsible Party: Principal Investigator, Gali Garmy, Dr Gali Garmi, HaEmek Medical Center, Israel
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 0056-17-EMC
Record Dates: First submitted 2017-09-04; First posted 2017-09-06 (Actual); Last update posted 2023-10-11 (Actual); Status verified 2023-10

CONDITIONS: Obstetric Labor; Pregnancy in Diabetics
Keywords: Gestational diabetes mellitus; Pre-gestational diabetes mellitus; Treatment; Neonatal hypoglycemia
MeSH Terms: conditions — Pregnancy in Diabetics; Diabetes, Gestational | interventions — Insulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- glucose solution and insulin (Active Comparator): Participants will receive intravenous saline solution boosted with 5% glucose + 8 units regular insulin in a rate of 125 mL/h.
  Interventions: Drug: glucose solution and Insulin; Drug: glucose solution only
- glucose solution only (Active Comparator): Participants will receive intravenous saline solution boosted with 5% glucose in a rate of 125 mL/h.
  Interventions: Drug: glucose solution and Insulin

INTERVENTIONS:
Drug: glucose solution and Insulin — Women in group 1, will receive intravenous saline solution boosted with 5% glucose combined with 8 units of insulin at a rate of 125mL/h. The desirable intrapartum glucose level will be 70 to 100 mg/dL. Glucose levels will be checked hourly.
  Glucose level between 100-140 mg/dL will be treated with additional intravenous insulin, 1 units/hour.
  Glucose level between 141-160 mg/dL will be treated with intravenous insulin, 2 units/hour. Additionally, the 5% glucose solution will be substitute with lactated Ringer's solution.
  Glucose level between 161-200 mg/dL will be treated with intravenous insulin, 4 units/hour.
  Glucose level above 200 mg/dL will be treated with intravenous insulin, 6 units/hour.
  Other Names: Group 1
Drug: glucose solution only — Women in group 2, will receive intravenous saline solution boosted with 5% glucose only, at a rate of 125mL/h. Women in this group will be treated similar to group 1 if glucose levels crossed over 100 mg/dL.
  Other Names: Group 2
  Arms: glucose solution and insulin

SUMMARY:
This study aims to examine the effect of intrapartum treatment of diabetic women with combined glucose and constant insulin infusion compared to glucose alone on the incidence of neonatal hypoglycemia. Pregnant women with diabetes in pregnancy will be randomly divided during labor to 2 groups: group 1, will receive intravenous glucose with constant insulin infusion; group 2 will receive intravenous glucose alone. The primary outcome is the incidence of neonatal hypoglycemia.

DETAILED DESCRIPTION:
About 2 to 9% of pregnant women are diagnosed with gestational diabetes. Peripartum complications attributed to diabetes include: birth trauma, neonatal hypoglycemia and hyperinsulinemia and neonatal hyperbilirubinemia. The incidence of neonatal hypoglycemia is about 40%. Strict glycemic control may lower the risk of neonatal complications. There is a lack of evidence on how to manage women with diabetes during labor. Previous studies recommended the use of intravenous saline solution boosted with 5% glucose and insulin as needed, glucose 5% with constant insulin infusion and others recommended the use lactated Ringer's solution. Most of these studies are either retrospective or have a small number of participants.

In this study we will examine the effect of 2 different protocols on glycemic control during labor and the immediate neonatal period. Women in group 1, will receive intravenous saline solution boosted with 5% glucose and constant insulin infusion. Women in group 2, will receive intravenous saline solution boosted with 5% glucose alone. The desirable intrapartum glucose level will be 70 to 100 mg/dL. Glucose levels will be checked hourly. Women in both groups will receive additional insulin infusion in cases of glucose levels above 100 mg/dL. Additionally, the 5% glucose solution will be substitute with lactated Ringer's solution in cases of glucose levels above 140 mg/dL.

Intravenous fluid regimens will be assigned according to a computer randomization sequence generation program. Women will randomly assigned to the 2 groups in a 1:1 ratio. The randomization sequence results will be kept in the delivery ward in a closed study box. Site investigators will enroll participants after confirming eligibility. The sequence will be concealed until intervention is assigned (and after obtaining a signed informed consent).

Our hypothesis is that 5% glucose combined with constant insulin infusion will achieve better glycemic control and thus will lead to lower rate of neonatal hypoglycemia. In order to detect a reduction of neonatal hypoglycemia from 40% to 20%, 182 women will be needed in both groups in order to achieve a level of significance of 95% (α, 2-sided = 0.05) and a power of 80% (β = 0.2).

ELIGIBILITY:
Inclusion Criteria:

* >37 weeks gestation
* gestational diabetes mellitus according to Carpenter and Coustan
* pregestational diabetes mellitus

Exclusion Criteria:

* Intrauterine fetal death
* estimated fetal weight<10p
* multiple gestation
* major fetal malformations

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2017-10-31 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Neonatal hypoglycemia | 2-3 hours postpartum
  about 2-3 hours postpartum the neonate will have a capillary glucose test

SECONDARY OUTCOMES:
Maternal glycemic control during labor | 24 hours
  During labor glucose level will be obtained every hour. Average glucose level during labor will be calculated after labor.
Maternal urine ketones | 1 hour
  Immediately post partum maternal urine will be checked for ketones
Total amount of regular insulin during labor | 24 hours
  The total amount of regular insulin during labor will be calculated post partum
Mode of delivery | 1 hour
  Mode of delivery
Length of delivery | 24 hours
  Length of delivery
Breastfeeding | 48 hours
  How many women breastfed in every study group
Neonatal APGAR score | 5 minutes
  Neonatal APGAR score
Umbilical cord PH | 30 minutes
  Umbilical cord PH
Umbilical cord glucose level | 30 minutes
  Umbilical cord glucose level
The need for neonatal IV glucose infusion | 48 hours
  The need for neonatal IV glucose infusion
Neonatal jaundice | 48 hours
  Neonatal jaundice- hyperbilirubinemia
Length of neonatal hospital stay | 30 days
  Length of neonatal hospital stay
NICU admission | 48 hours
  NICU admission

CONTACTS AND LOCATIONS:
Overall Officials: Gali Gali, MD, Principal Investigator — HaEmemk Medical Center, Afula, Israel.
Locations (1):
- HaEmek medical center, Afula, Israel

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Soler NG, Soler SM, Malins JM. Neonatal morbidity among infants of diabetic mothers. Diabetes Care. 1978 Nov-Dec;1(6):340-50. doi: 10.2337/diacare.1.6.340. PMID 729447
- [Background] Sacks DA, Hadden DR, Maresh M, Deerochanawong C, Dyer AR, Metzger BE, Lowe LP, Coustan DR, Hod M, Oats JJ, Persson B, Trimble ER; HAPO Study Cooperative Research Group. Frequency of gestational diabetes mellitus at collaborating centers based on IADPSG consensus panel-recommended criteria: the Hyperglycemia and Adverse Pregnancy Outcome (HAPO) Study. Diabetes Care. 2012 Mar;35(3):526-8. doi: 10.2337/dc11-1641. PMID 22355019
- [Background] Taricco E, Radaelli T, Rossi G, Nobile de Santis MS, Bulfamante GP, Avagliano L, Cetin I. Effects of gestational diabetes on fetal oxygen and glucose levels in vivo. BJOG. 2009 Dec;116(13):1729-35. doi: 10.1111/j.1471-0528.2009.02341.x. Epub 2009 Oct 13. PMID 19832834
- [Background] HAPO Study Cooperative Research Group; Metzger BE, Lowe LP, Dyer AR, Trimble ER, Chaovarindr U, Coustan DR, Hadden DR, McCance DR, Hod M, McIntyre HD, Oats JJ, Persson B, Rogers MS, Sacks DA. Hyperglycemia and adverse pregnancy outcomes. N Engl J Med. 2008 May 8;358(19):1991-2002. doi: 10.1056/NEJMoa0707943. PMID 18463375
- [Background] Reece EA, Leguizamon G, Wiznitzer A. Gestational diabetes: the need for a common ground. Lancet. 2009 May 23;373(9677):1789-97. doi: 10.1016/S0140-6736(09)60515-8. PMID 19465234
- [Background] Ju H, Rumbold AR, Willson KJ, Crowther CA. Borderline gestational diabetes mellitus and pregnancy outcomes. BMC Pregnancy Childbirth. 2008 Jul 30;8:31. doi: 10.1186/1471-2393-8-31. PMID 18664297
- [Background] Catalano PM, McIntyre HD, Cruickshank JK, McCance DR, Dyer AR, Metzger BE, Lowe LP, Trimble ER, Coustan DR, Hadden DR, Persson B, Hod M, Oats JJ; HAPO Study Cooperative Research Group. The hyperglycemia and adverse pregnancy outcome study: associations of GDM and obesity with pregnancy outcomes. Diabetes Care. 2012 Apr;35(4):780-6. doi: 10.2337/dc11-1790. Epub 2012 Feb 22. PMID 22357187
- [Background] Committee on Fetus and Newborn; Adamkin DH. Postnatal glucose homeostasis in late-preterm and term infants. Pediatrics. 2011 Mar;127(3):575-9. doi: 10.1542/peds.2010-3851. Epub 2011 Feb 28. PMID 21357346
- [Result] Carron Brown S, Kyne-Grzebalski D, Mwangi B, Taylor R. Effect of management policy upon 120 Type 1 diabetic pregnancies: policy decisions in practice. Diabet Med. 1999 Jul;16(7):573-8. doi: 10.1046/j.1464-5491.1999.00124.x. PMID 10445833
- [Result] Kline GA, Edwards A. Antepartum and intra-partum insulin management of type 1 and type 2 diabetic women: Impact on clinically significant neonatal hypoglycemia. Diabetes Res Clin Pract. 2007 Aug;77(2):223-30. doi: 10.1016/j.diabres.2006.10.024. Epub 2006 Nov 28. PMID 17126946
- [Result] Lean ME, Pearson DW, Sutherland HW. Insulin management during labour and delivery in mothers with diabetes. Diabet Med. 1990 Feb;7(2):162-4. doi: 10.1111/j.1464-5491.1990.tb01352.x. PMID 2137758
- [Result] Balsells M, Corcoy R, Adelantado JM, Garcia-Patterson A, Altirriba O, de Leiva A. Gestational diabetes mellitus: metabolic control during labour. Diabetes Nutr Metab. 2000 Oct;13(5):257-62. PMID 11105967
- [Result] Hussain K, Sharief N. The inaccuracy of venous and capillary blood glucose measurement using reagent strips in the newborn period and the effect of haematocrit. Early Hum Dev. 2000 Feb;57(2):111-21. doi: 10.1016/s0378-3782(99)00060-2. PMID 10735458
- [Result] Hernandez-Rivas E, Flores-Le Roux JA, Benaiges D, Sagarra E, Chillaron JJ, Paya A, Puig-de Dou J, Goday A, Lopez-Vilchez MA, Pedro-Botet J. Gestational diabetes in a multiethnic population of Spain: clinical characteristics and perinatal outcomes. Diabetes Res Clin Pract. 2013 May;100(2):215-21. doi: 10.1016/j.diabres.2013.01.030. Epub 2013 Mar 26. PMID 23538268
- [Result] Carpenter MW, Coustan DR. Criteria for screening tests for gestational diabetes. Am J Obstet Gynecol. 1982 Dec 1;144(7):768-73. doi: 10.1016/0002-9378(82)90349-0. PMID 7148898